CLINICAL TRIAL: NCT02419495
Title: Phase IB Study to Evaluate the Safety of Selinexor (KPT-330) in Combination With Multiple Standard Chemotherapy or Immunotherapy Agents in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively Complete
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0640; NCI-2015-00693 (Registry Identifier: NCI-Clinical Trial Registry); 2014-0640 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2024-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Fallopian Tube Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Renal Cell Carcinoma; Ovarian Carcinoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Primary Peritoneal Carcinoma; Stage III Lung Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Triple-Negative Breast Carcinoma; Unresectable Lung Non-Small Cell Carcinoma; Unresectable Melanoma; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Melanoma; Carcinoma, Renal Cell; Ovarian Neoplasms; Lung Neoplasms; Triple Negative Breast Neoplasms | interventions — Capecitabine; Carboplatin; Cyclophosphamide; Doxorubicin; eribulin; Fluorouracil; dehydroftorafur; Ipilimumab; CTLA-4 Antigen; Irinotecan; Leucovorin; Nivolumab; olaparib; Oxaliplatin; Paclitaxel; Taxes; pembrolizumab; Pemetrexed; selinexor; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Arm A (selinexor, carboplatin) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8, and 15 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Carboplatin; Drug: Selinexor
- Arm B (selinexor, paclitaxel) (Experimental): Patients receive selinexor PO twice weekly (e.g. Monday/Wednesday or Tuesday/Thursday or Wednesday/Friday or Thursday/Saturday or Friday/Sunday) on days 1-14. Patients then receive selinexor PO on days 1, 3, 8 and 10 and paclitaxel IV over 3 hours on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. After 8 cycles of combination treatment, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Paclitaxel; Drug: Selinexor
- Arm C (selinexor, eribulin) (Experimental): Patients receive selinexor PO on days 1, 8, and 15 and eribulin IV over 1 hour on days 1 and 8. Combination treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Eribulin; Drug: Selinexor
- Arm D (selinexor, doxorubicin, cyclophosphamide) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8, and 15, doxorubicin IV over 90 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Selinexor
- Arm E (selinexor, carboplatin, paclitaxel) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8, and 15 and carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment repeats every 21 days for up to 8 cycles depending con cancer type (6 cycles for non-small cell lung cancer, up to 8 cycles for ovarian cancer and other histological malignancies) in the absence of disease progression or unacceptable toxicity. After 6 to 8 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Selinexor
- Arm F (selinexor, carboplatin, pemetrexed) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8, and 15 and carboplatin IV over 30 minutes and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Selinexor
- Arm G (selinexor, topotecan hydrochloride) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8, and 15 and topotecan hydrochloride IV over 30 minutes on days 1-5. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. After 8 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Selinexor; Drug: Topotecan
- Arm H (selinexor, FOLFIRI) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8, 15 and 22, irinotecan hydrochloride IV over 90 minutes, fluorouracil IV continuously over 48 hours and leucovorin calcium IV over 2 hours on days 1 and 15. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Selinexor
- Arm I (selinexor, irinotecan hydrochloride) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8 and 15 and irinotecan hydrochloride IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. After 8 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Irinotecan Hydrochloride; Drug: Selinexor
- Arm J (selinexor, capecitabine, oxaliplatin) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8 and 15, capecitabine PO twice daily (BID) on days 1-14 and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. After 8 cycles, patients can continue single agent selinexor until disease progression.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Selinexor
- Arm K (selinexor, olaparib) (ARM CLOSED) (Experimental): Patients receive selinexor PO on days 1, 8, 15, and 22 and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib; Drug: Selinexor
- Arm L (selinexor, pembrolizumab) (Experimental): Patients receive selinexor PO twice weekly (e.g. Monday/Wednesday or Tuesday/Thursday or Wednesday/Friday or Thursday/Saturday or Friday/Sunday) and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Selinexor
- Arm M (selinexor, nivolumab (Experimental): Patients receive selinexor PO twice weekly (e.g. Monday/Wednesday or Tuesday/Thursday or Wednesday/Friday or Thursday/Saturday or Friday/Sunday) and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Selinexor
- Arm P (selinexor, nivolumab, ipilimumab) (Experimental): Patients receive selinexor PO on days 1, 8, 15, 22, 29, and 36, nivolumab IV over 30 minutes on days 1, 15, and 29, and ipilimumab PO QD on day 1. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Drug: Selinexor
- Arms N and O (selinexor, nivolumab, ipilimumab) (Experimental): Patients receive selinexor PO on days 1, 8, and 15, nivolumab IV over 30 minutes on day 1, and ipilimumab PO QD on day 1. Cycles repeat every 3 weeks for 4 cycles. Starting cycle 5, patients receive selinexor PO on days 1, 8, 15, and 22 and nivolumab IV over 30 minutes on day 1. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Drug: Selinexor

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Arm J (selinexor, capecitabine, oxaliplatin) (ARM CLOSED)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm A (selinexor, carboplatin) (ARM CLOSED); Arm E (selinexor, carboplatin, paclitaxel) (ARM CLOSED); Arm F (selinexor, carboplatin, pemetrexed) (ARM CLOSED)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm D (selinexor, doxorubicin, cyclophosphamide) (ARM CLOSED)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Arm D (selinexor, doxorubicin, cyclophosphamide) (ARM CLOSED)
Drug: Eribulin — Given IV
  Other Names: ER-086526
  Arms: Arm C (selinexor, eribulin)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm H (selinexor, FOLFIRI) (ARM CLOSED)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm P (selinexor, nivolumab, ipilimumab); Arms N and O (selinexor, nivolumab, ipilimumab)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
  Arms: Arm H (selinexor, FOLFIRI) (ARM CLOSED); Arm I (selinexor, irinotecan hydrochloride) (ARM CLOSED)
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm H (selinexor, FOLFIRI) (ARM CLOSED)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
  Arms: Arm M (selinexor, nivolumab; Arm P (selinexor, nivolumab, ipilimumab); Arms N and O (selinexor, nivolumab, ipilimumab)
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
  Arms: Arm K (selinexor, olaparib) (ARM CLOSED)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
  Arms: Arm J (selinexor, capecitabine, oxaliplatin) (ARM CLOSED)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm B (selinexor, paclitaxel); Arm E (selinexor, carboplatin, paclitaxel) (ARM CLOSED)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm L (selinexor, pembrolizumab)
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: Arm F (selinexor, carboplatin, pemetrexed) (ARM CLOSED)
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
  Arms: Arm G (selinexor, topotecan hydrochloride) (ARM CLOSED)

SUMMARY:
This phase Ib trial studies the side effects and best dose of selinexor when given together with several different standard chemotherapy or immunotherapy regimens in treating patients with malignancies that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Selinexor may stop the growth of cancer cells by blocking enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Studying selinexor with different standard chemotherapy or immunotherapy regimens may help doctors learn the side effects and best dose of selinexor that can be given with different types of treatments in one study.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the safety and tolerability of selinexor when given in combination with standard chemotherapy or immunotherapy regimens.

SECONDARY OBJECTIVE:

I. To determine disease control rate, objective tumor response rate, and progression free survival of selinexor administered with standard chemotherapy or immunotherapy treatments.

EXPLORATORY OBJECTIVES:

I. To determine the correlation of translational biomarkers. II. To compare serial assessment of mutation status in biopsies obtained at baseline and progression after clinical response to combination therapy.

III. To assess the efficacy of olanzapine as incorporated in the National Comprehensive Cancer Network (NCCN) guidelines for the management of chemotherapy-induced nausea and cachexia.

OUTLINE: This is a dose-escalation study of selinexor. Patients are assigned to 1 of 15 treatment arms.

ARM A: Patients receive selinexor orally (PO) on days 1, 8, and 15 and carboplatin intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM B: Patients receive selinexor PO twice weekly (e.g. Monday/Wednesday or Tuesday/Thursday or Wednesday/Friday or Thursday/Saturday or Friday/Sunday) on days 1-14. Patients then receive selinexor PO on days 1, 3, 8 and 10 and paclitaxel IV over 3 hours on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. After 8 cycles, of combination treatment, patients can continue single agent selinexor until disease progression.

ARM C: Patients receive selinexor PO on days 1, 8, and 15 and eribulin IV over 1 hour on days 1 and 8. Combination treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression.

ARM D: Patients receive selinexor PO on days 1, 8, and 15, doxorubicin IV over 90 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM E: Patients receive selinexor PO on days 1, 8, and 15 and carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Treatment repeats every 21 days for up to 8 cycles depending on cancer type (6 cycles for non-small cell lung cancer, up to 8 cycles for ovarian cancer and other histological malignancies) in the absence of disease progression or unacceptable toxicity. After 6 to 8 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM F: Patients receive selinexor PO on days 1, 8, and 15 and carboplatin IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM G: Patients receive selinexor PO on days 1, 8, and 15 and topotecan IV over 30 minutes on days 1-5. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. After 8 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM H: Patients receive selinexor PO on days 1, 8, 15 and 22, irinotecan hydrochloride IV over 90 minutes, fluorouracil continuous IV and leucovorin calcium IV over 2 hours on days 1 and 15. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 6 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM I: Patients receive selinexor PO on days 1, 8 and 15 and irinotecan hydrochloride IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. After 8 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM J: Patients receive selinexor PO on days 1, 8 and 15, capecitabine PO twice daily (BID) on days 1-14 and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. After 8 cycles, patients can continue single agent selinexor until disease progression. (ARM CLOSED)

ARM K: Patients receive selinexor PO on days 1, 8, 15, and 22 and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. (ARM CLOSED)

ARM L: Patients receive selinexor PO twice weekly (e.g. Monday/Wednesday or Tuesday/Thursday or Wednesday/Friday or Thursday/Saturday or Friday/Sunday) and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM M: Patients receive selinexor PO twice weekly (e.g. Monday/Wednesday or Tuesday/Thursday or Wednesday/Friday or Thursday/Saturday or Friday/Sunday) and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARMS N AND O: Patients receive selinexor PO on days 1, 8, and 15, nivolumab IV over 30 minutes on day 1, and ipilimumab PO QD on day 1. Cycles repeat every 3 weeks for 4 cycles. Starting cycle 5, patients receive selinexor PO on days 1, 8, 15, and 22 and nivolumab IV over 30 minutes on day 1. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM P: Patients receive selinexor PO on days 1, 8, 15, 22, 29, and 36, nivolumab IV over 30 minutes on days 1, 15, and 29, and ipilimumab PO QD on day 1. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients may continue to receive selinexor and chemotherapy after confirmed progressive disease in the absence of clinical deterioration and if the investigator considers that the patient continues to receive benefit from the treatment.

After completion of study treatment, patients are followed up every 12 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant neoplasms (not including hematological malignancies and brain tumors) untreated or previously treated requiring further treatment; patients in Arm L (pembrolizumab), Arm M (nivolumab), and Arms N, O, P (nivolumab and ipilimumab) that have Food and Drug Administration (FDA)-approved indications for nivolumab, ipilimumab, and pembrolizumab do not have to fail first line nivolumab, ipilimumab, or pembrolizumab, and these patients may be treatment naïve if they have disease where pembrolizumab or nivolumab are FDA approved for the first-line setting
* For all arms except Arm L (pembrolizumab), Arm M (nivolumab), and Arms N, O, P (nivolumab and ipilimumab) patients must have failed prior standard curative chemotherapy for their disease; subjects must have failed, be intolerant to, or be ineligible for any potentially curative approved treatment, irrespective of line of therapy
* Patients must have measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* The patient must be recovered from a prior major surgery; the major surgery must be performed at least 4 weeks prior to consent date
* Platelets >= 125 x 10^9/L (For Arm L pembrolizumab, Arm M nivolumab and Arms N, O, P [nivolumab and ipilimumab] and expansion cohorts for all arms, platelets >= 100 x 10^9/L)
* Hemoglobin >= 10 g/dL (For Arm L pembrolizumab, Arm M nivolumab and Arms N, O, P [nivolumab and ipilimumab] and expansion cohorts for all arms, hemoglobin >= 9 g/dL)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (For Arm L pembrolizumab, Arm M nivolumab and Arms N, O, P [nivolumab and ipilimumab], ANC >= 1.0 x 10^9/L)
* Transfusions and growth factors are allowed
* Alanine transaminase (alanine aminotransferase [ALT]) =< 2 x upper normal limit (ULN) (in the expansion cohort, patients with known liver involvement may have ALT =< 5 x ULN); aspartate aminotransferase (AST) =< 2 x ULN (in the expansion cohort, patients with known liver involvement may have AST =< 5 x ULN)
* Alkaline phosphatase < 4 x ULN
* Total bilirubin =< 2 x ULN (in the expansion cohort, patients with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must have a total bilirubin of =< 3 x ULN)
* Renal function defined as a calculated or measured glomerular filtration rate (GFR) >= 30 mL/min. For patients with renal cell carcinoma (RCC), the GFR may be defined as >= 25 mL/min
* The patient has recovered to grade =< 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03 (NCI-CTCAE v4.03) from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies, with the exception of alopecia; the exceptions for such effects are allowed lab values of =< grade 2 specified elsewhere in these inclusion criteria
* Life expectancy of at least 12 weeks
* Able to swallow and retain oral medication
* Patients must give informed consent according to the rules and regulations of the individual participating sites
* Negative serum pregnancy test in women of childbearing potential within 7 days of first dose of treatment and patients of child-bearing potential must agree to use effective contraception during/after 3 months post dose; a woman of childbearing potential is defined as a premenopausal female capable of becoming pregnant; this includes women on oral, injectable or mechanical contraception; women who are single and women whose male sexual partners have been vasectomized or whose male sexual partners have received or are utilizing mechanical contraceptive devices
* For the Arm B (paclitaxel) expansion cohort, patients must have ovarian carcinoma, fallopian tube, or peritonea carcinoma
* For Arm C (eribulin) expansion cohort, patients must have triple negative breast cancer (eribulin naive)
* For Arm M (nivolumab) expansion phase, patients must have biopsiable disease
* For the Arm N (nivolumab and ipilimumab), patients must have metastatic or unresectable renal cell carcinoma (RCC)
* For the Arm O (nivolumab and ipilimumab) escalation and expansion Cohort O-1, patients must have metastatic or unresectable melanoma
* For the Arm O (nivolumab and ipilimumab) expansion Cohort O-2, patients must have metastatic or advanced solid tumors (non-melanoma, non-renal cell carcinoma, or non- non-small cell lung carcinoma)
* For the Arm P (nivolumab and ipilimumab), patients must have metastatic or unresectable non-small cell lung carcinoma (NSCLC)

Exclusion Criteria:

* Evidence of complete or partial bowel obstruction
* Patients with primary central nervous system (CNS) tumor or CNS tumor involvement; however, patients with metastatic CNS tumors may participate in this study if the patient is:

  * > 4 weeks from prior therapy completion (including radiation and/or surgery)
  * Clinically stable with respect to the CNS tumor at the time of study entry
  * Not receiving steroid therapy in treating CNS tumor or CNS tumor involvement
  * Not receiving anti-convulsive medications (that were started for brain metastases)
* Need of total parenteral nutrition
* Prior treatment with an agent targeting the exportin
* Allergic to selinexor or any of the chemotherapy intended to receive
* Pregnancy or lactation
* Radiation (except planned or ongoing palliative radiation to bone outside of the region of measurable disease) =< 3 weeks prior to study drug administration date
* Chemotherapy, or immunotherapy or any other systemic anticancer therapy =< 3 weeks prior to study drug administration date; patients receiving anti-PD-1 treatment, and continue to receiving this treatment in combination with selinexor (Arms L, M, N, O, and P), can start receiving the selinexor and anti-PD-1 combination without washout of the prior anti-PD-1 antibody
* Diagnosis or recurrence of invasive cancer other than the present cancer within 3 years (except basal or squamous cell carcinoma of the skin that has been definitively treated)
* Major surgery within four weeks before consent date
* Unstable cardiovascular function: symptomatic ischemia (chest pain of cardiac origin), or uncontrolled clinically significant conduction abnormalities (e.g. ventricular tachycardia on antiarrhythmics are excluded and 1st degree atrioventricular [AV] block or asymptomatic left anterior fascicular block [LAFB]/right bundle branch block [RBBB] will not be excluded), or congestive heart failure (CHF) of New York Heart Association (NYHA) class >= 3, or myocardial infarction (MI) within 3 months of consent date
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to the first dose; active infection with concurrent treatment is acceptable only if the patient is clinically stable
* Significantly diseased (as determined by the principal investigator [PI] or treating physician) or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea
* Treatment with an investigational anti-cancer study drug within 3 weeks prior to study drug administration date
* Concurrent therapy with approved or investigational anticancer therapeutics
* Medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Men whose partner is a woman of child-bearing potential, (i.e. biologically able to conceive), and who is not employing two forms of highly effective contraception; highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 3 months after the end of study treatment; women of child-bearing potential is defined as sexually mature women who are not surgically sterile or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months)
* For Arms L (pembrolizumab) and M (nivolumab), and Arms N, O, P (nivolumab and ipilimumab), subjects with an active, known or suspected autoimmune disease; subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* For Arms L (pembrolizumab) and M (nivolumab), and Arms N, O, P (nivolumab and ipilimumab), subjects receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or other form of immunosuppressive therapy within 7 days before the first dose of study treatment; use of inhaled or topical steroids or systemic corticosteroids =< 10 mg is permitted; in addition, physiologic steroid replacement with hydrocortisone is allowed
* For Arms L (pembrolizumab) and M (nivolumab), and Arms N, O, P (nivolumab and ipilimumab), history of a prior grade 3 or 4 immune-related adverse event (irAE) or any grade ocular irAE from prior immunotherapy
* For the Arm O (nivolumab and ipilimumab) expansion Cohort O-2, patients must not have melanoma, RCC, or NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

SECONDARY OUTCOMES:
Disease control rate (complete response, partial response + stable disease for at least 6 months | Up to 3 years
  Assessed according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria). Estimated separately for each cohort with appropriate 95% confidence intervals.
Objective tumor response rate (complete response + partial response) | Up to 3 years
  Assessed according to RECIST 1.1 criteria. Estimated separately for each cohort with appropriate 95% confidence intervals.
Progression-free survival (PFS) | The time between the course 1 start date and the date of disease progression or death, whichever is reported first, assessed up to 3 years
  PFS distribution will be estimated using the Kaplan-Meier product limit method and summary measures such as the median value and probabilities will be reported at selected times (with appropriate 95% confidence intervals).
Overall survival (OS) | Up to 3 years
  OS distribution will be estimated using the Kaplan-Meier product limit method and summary measures such as the median value and probabilities will be reported at selected times (with appropriate 95% confidence intervals).
Incidence of adverse events | Up to 3 years
  Will be graded according to NCI CTCAE version 4.03.

OTHER OUTCOMES:
Serial mutations in biopsies | Up to 30 days after last dose of treatment
Severity of nausea and vomiting | Up to 3 years
Change in weight | Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- [Derived] Alhalabi O, Gouda MA, Milton DR, Momin HA, Yilmaz B, Stephen B, Ejezie CL, Moyers JT, Gurses SA, How J, Fu S, Rodon J, Hong DS, Piha-Paul SA, Subbiah V, Elena Dumbrava E, Karp DD, Janku F, Meric-Bernstam F, Tannir NM, Naing A. A Phase IB Trial of Selinexor in Combination With Immune Checkpoint Blockade in Patients With Advanced Renal Cell Carcinoma. Cancer Med. 2025 Feb;14(4):e70280. doi: 10.1002/cam4.70280. PMID 39945382
- [Derived] Gouda MA, Zarifa A, Yang Y, Stephen B, Gurses SA, Sprenger A, Tian Y, Derbala MH, Oliva IG, Meric-Bernstam F, Patel SP. Selinexor (KPT-330) in Combination with Immune Checkpoint Inhibition in Uveal Melanoma: A Phase 1B Trial. J Immunother Precis Oncol. 2025 Jan 15;8(1):82-88. doi: 10.36401/JIPO-24-10. eCollection 2025 Feb. PMID 39816915
- [Derived] Altan M, Tu J, Milton DR, Yilmaz B, Tian Y, Fossella FV, Mott FE, Blumenschein GR, Stephen B, Karp DD, Meric-Bernstam F, Heymach JV, Naing A. Safety, tolerability, and clinical activity of selinexor in combination with pembrolizumab in treatment of metastatic non-small cell lung cancer. Cancer. 2023 Sep 1;129(17):2685-2693. doi: 10.1002/cncr.34820. Epub 2023 May 2. PMID 37129197
- [Derived] Thein KZ, Piha-Paul SA, Tsimberidou A, Karp DD, Janku F, Fu S, Subbiah V, Hong DS, Yap TA, Shah J, Milton DR, McQuinn L, Gong J, Tran Y, Carter BW, Colen R, Meric-Bernstam F, Naing A. Selinexor in combination with standard chemotherapy in patients with advanced or metastatic solid tumors. Exp Hematol Oncol. 2021 Dec 29;10(1):59. doi: 10.1186/s40164-021-00251-0. PMID 34965890
- [Derived] Thein KZ, Karp DD, Tsimberidou A, Gong J, Sulovic S, Shah J, Milton DR, Hong DS, Janku F, McQuinn L, Stephen BA, Colen R, Carter BW, Yap TA, Piha-Paul SA, Fu S, Meric-Bernstam F, Naing A. Selinexor in combination with carboplatin and paclitaxel in patients with advanced solid tumors: Results of a single-center, multi-arm phase Ib study. Invest New Drugs. 2022 Apr;40(2):290-299. doi: 10.1007/s10637-021-01188-1. Epub 2021 Sep 25. PMID 34562230
- [Derived] Thein KZ, Piha-Paul SA, Tsimberidou A, Karp DD, Janku F, Zarifa A, Shah J, Milton DR, Bean S, McQuinn L, Gong J, Colen R, Carter BW, Subbiah V, Ogbonna DC, Pant S, Meric-Bernstam F, Naing A. Selinexor in combination with topotecan in patients with advanced or metastatic solid tumors: Results of an open-label, single-center, multi-arm phase Ib study. Invest New Drugs. 2021 Oct;39(5):1357-1365. doi: 10.1007/s10637-021-01119-0. Epub 2021 Apr 28. PMID 33909232
- See also: M D Anderson Cancer Center — http://www.mdanderson.org